CLINICAL TRIAL: NCT05105204
Title: ArteVu Blood Pressure Accuracy Study
Acronym: ARTEVU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cardio Ring Technologies, Inc. Taiwan Branch (Industry)
Collaborators: Taipei Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: N202106030
Record Dates: First submitted 2021-10-04; First posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Blood Pressure
Keywords: non-invasive blood pressure monitor; arterial waveform

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Individuals need intra-arterial catheter at the radial artery for blood pressure monitoring: Individuals who requiring the use of intra-arterial catheter at the radial artery for continuous blood pressure monitoring for at least two hours as part of their planned care.
  Interventions: Device: ArteVu

INTERVENTIONS:
Device: ArteVu — The study participants will concurrently undergo noninvasive blood pressure monitoring with the ArteVu finger clip applied to the same extremity that is being used to measure the radial artery pressure.

SUMMARY:
A continuous noninvasive blood pressure monitoring digital fingertip clip device, the ArteVu, will be compared against the reference arterial catheter during operation. The device safety and its blood pressure accuracy will be examined in the study.

DETAILED DESCRIPTION:
ArteVu is a non-invasive and continuous blood pressure monitor. It detects the arterial pressure waveform with a force sensor that detects the arterial pulsation that produces changes in pressure transmitted through the subcutaneous tissue overlying or adjacent to the digital arteries. The data is transmitted to a parameter module to display noninvasive and continuous blood pressure in a hospital setting. The primary objective of this study is to validate ArteVu's blood pressure and heart rate measurement accuracy by comparing its values simultaneously with the corresponding values obtained from an invasive radial arterial line. The secondary objective is to evaluate the effectiveness of utilizing ArteVu for continuous blood pressure measurements. The study population includes 50 patients undergoing surgery who requires general anesthesia and continuous blood pressure measurement with a radial arterial line. Blood pressure values measured from the arterial line will be recorded simultaneously during ArteVu's measurements.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 20 years
2. Requiring general anesthesia and continuous blood pressure measurement with a radial arterial line
3. Limb circumference is within 22 cm - 32 cm
4. The width of the first knuckle of the index/middle/Ring finger is less than 19.8 mm
5. Ease of access to the finger and arm used for ArteVu
6. Able to provide written informed consent for participation in the study

Exclusion Criteria:

1. Pregnant patients
2. Medical or surgical condition that prevents the ability to apply the ArteVu device on an upper extremity finger or the ipsilateral arm such as impaired skin integrity
3. Operations involving the upper extremities or the blood vessels of the upper extremities
4. Arthritis or severe deformities of the hand and fingers
5. Prosthetic devices or jewelry that cannot be removed from the finger or the ipsilateral arm to be used for the ArteVu device
6. History of malignant hyperthermia
7. Raynaud's disease affecting the fingers or hands
8. Topical allergy to Acrylonitrile Butadiene Styrene(ABS), Polycarbonate(PC), or silicone
9. Swelling, edema or lymphedema of the upper extremity
10. Participants with upper extremity occlusive peripheral vascular diseases
11. Inability of the patient to provide written informed consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient enrollment will continue until at least 30% are male; 30% are female; at least 40 % patients have a limb circumference that lies within the upper half of 22-32 cm; at least 40 % are within the lower half of 22-32 cm; in addition, 50 complete one-hour CNBP and NBP data sets are obtained. To assure that a sufficient range of blood pressure values are obtained, at least 10% of the measurements shall have invasive reference systolic blood pressure(SBP) lower or equal to 100 mmHg. At least 10% of the measurements shall have invasive reference SBP higher or equal to 160 mmHg. At least 10% of the measurements shall have invasive reference diastolic blood pressure(DBP) lower or equal to 70mmHg. At least 10% of the measurements shall have invasive reference DBP higher or equal to 85 mmHg.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-09-14 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Blood pressure and heart rate measurement accuracy | around two hours.
  To validate ArteVu's blood pressure and heart rate measurement accuracy by comparing its values simultaneously with the corresponding values obtained intra-arterially from an invasive radial arterial line, meeting a bias (as measured by overall mean difference) less than 5 mmHg and a standard deviation less than 8 mmHg for systolic and diastolic blood pressure. This accuracy satisfies the limits established for the validation of automatic blood pressure measurement according to the ANSI/AAMI/ISO 81060-2 standard.

CONTACTS AND LOCATIONS:
Overall Officials: Chuen-Chau Chang, M.D,PhD., Principal Investigator — Taipei Medical University Hospital
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
IPD (study protocol and analytic code) that underlines the results reported in a further publication article, after de-identification.
Supporting Information: Study Protocol, Analytic Code
Time Frame: The estimated study completion date is 2022-6-30. These supporting information would become available beginning 3 months and ending 5 years following article publication.
Access Criteria: Researches who provide a methodologically sound proposal.

REFERENCES:
- [Background] Williams JS, Brown SM, Conlin PR. Videos in clinical medicine. Blood-pressure measurement. N Engl J Med. 2009 Jan 29;360(5):e6. doi: 10.1056/NEJMvcm0800157. No abstract available. PMID 19179309
- [Background] Stenglova A, Benes J. Continuous Non-Invasive Arterial Pressure Assessment during Surgery to Improve Outcome. Front Med (Lausanne). 2017 Nov 17;4:202. doi: 10.3389/fmed.2017.00202. eCollection 2017. PMID 29204425
- [Background] Froehler MT, Chitale R, Magarik JA, Fusco MR. Comparison of a pressure-sensing sheath and radial arterial line for intraoperative blood pressure monitoring in neurointerventional procedures. J Neurointerv Surg. 2018 Aug;10(8):784-787. doi: 10.1136/neurintsurg-2018-013769. Epub 2018 Feb 27. PMID 29487193
- [Background] Bland JM, Altman DG. Statistical methods for assessing agreement between two methods of clinical measurement. Lancet. 1986 Feb 8;1(8476):307-10. PMID 2868172
- [Background] Martina JR, Westerhof BE, van Goudoever J, de Beaumont EM, Truijen J, Kim YS, Immink RV, Jobsis DA, Hollmann MW, Lahpor JR, de Mol BA, van Lieshout JJ. Noninvasive continuous arterial blood pressure monitoring with Nexfin(R). Anesthesiology. 2012 May;116(5):1092-103. doi: 10.1097/ALN.0b013e31824f94ed. PMID 22415387
- [Background] Gratz I, Deal E, Spitz F, Baruch M, Allen IE, Seaman JE, Pukenas E, Jean S. Continuous Non-invasive finger cuff CareTaker(R) comparable to invasive intra-arterial pressure in patients undergoing major intra-abdominal surgery. BMC Anesthesiol. 2017 Mar 21;17(1):48. doi: 10.1186/s12871-017-0337-z. PMID 28327093
- [Background] Hohn A, Defosse JM, Becker S, Steffen C, Wappler F, Sakka SG. Non-invasive continuous arterial pressure monitoring with Nexfin does not sufficiently replace invasive measurements in critically ill patients. Br J Anaesth. 2013 Aug;111(2):178-84. doi: 10.1093/bja/aet023. Epub 2013 Mar 13. PMID 23485882
- [Background] Kim SH, Lilot M, Sidhu KS, Rinehart J, Yu Z, Canales C, Cannesson M. Accuracy and precision of continuous noninvasive arterial pressure monitoring compared with invasive arterial pressure: a systematic review and meta-analysis. Anesthesiology. 2014 May;120(5):1080-97. doi: 10.1097/ALN.0000000000000226. PMID 24637618
- [Result] Gerlach G, Hofer HW. Interaction of immobilized phosphofructokinase with soluble muscle proteins. Biochim Biophys Acta. 1986 May 2;881(3):398-404. doi: 10.1016/0304-4165(86)90032-2. PMID 2938635
- See also: Association for the Advancement of Medical Instrumentation. Non-invasive sphygmomanometers-Part 2: Clinical investigation of intermittent automated measurement type. This is also a results reference. — https://www.iso.org/standard/73339.html